CLINICAL TRIAL: NCT02881970
Title: Neonatal Hypoxic Ischemic Encephalopathy : Safety and Feasibility Study of a Curative Treatment With Autologous Cord Blood Stem Cells
Acronym: NEOSTEM
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-A01018-37; 2013-32 (Other: AP HM)
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Neonatal Hypoxic-ischaemic Encephalopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neonatal hypoxic-ischaemic encephalopathy (Experimental)
  Interventions: Drug: autologous cord blood stem cell

INTERVENTIONS:
Drug: autologous cord blood stem cell — Injection of 5.107 / kg autologous mononuclear cells from umbilical cord blood

SUMMARY:
Neonatal hypoxic-ischaemic encephalopathy is a dramatic perinatal complication due to brain asphyxia. Neurological and neurosensory sequelae are frequent in survivors, due to neuronal damage and loss.

Currently, only total or partial body hypothermia can partially prevent cell loss. However, no treatment exists to restore neuronal functions.

Cord blood stem cells are a promising treatment for the near future.

The primary objective of this study is to test the safety and feasibility of a curative treatment with autologous cord blood stem cell in neonatal hypoxic-ischaemic encephalopathy.

The secondary objectives are to test the efficacy of this curative treatment with cell with neurogenic potential on the prevention of neurologic sequelae, as well as to test the optimum timing of cell preparation administration

ELIGIBILITY:
Inclusion Criteria:

Term ≥ 36 weeks of gestation

* and (2) :
* a blood pH < 7 with base deficit > 12 mmol/l (at birth or within 60 minutes of age)
* or a blood pH between 7,01 and 7,15, with additionnal criteria:
* a history of acute perinatal event (e.g : abnormal fetal cardiac rate, cord prolapse, uterine rupture, maternal hemorrhage)
* and a 5 minutes Apgar score ≤ 5, or a continued need for resuscitation, including endotracheal or mask ventilation at 5 min after birth.
* signs of encephalopathy within 12 hours of age (Sarnat and Sarnat classification, score ≥ 2)
* ± abnormal electroencephalogram or aEEG within 12 hours of age
* therapeutic hypothermia.
* no maternal infection with VIH, HTLV 1 or 2, Hepatitis B or C virus.
* maternal negative serology for syphilis
* written parental consent

Exclusion Criteria:

* presence of known chromosomal anomaly.
* presence of major congenital anomalies. severe intrauterine growth restriction (weight <1800g)
* infants in extremis for whom no additional intensive therapy will be offered by attending neonatologist.

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2020-02-05 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Adverse clinical or paraclinical event rates due to stem cell preparation | 2years

SECONDARY OUTCOMES:
- Preliminary efficacy as measured by neurodevelopmental function | 2years

CONTACTS AND LOCATIONS:
Overall Officials: CATHERINE GEINDRE, Study Director — AP HM
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No